CLINICAL TRIAL: NCT03662750
Title: TSPO PET as a Measure of Post-stroke Brain Inflammation: a Natural History Cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Biogen (Industry); Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GBR-TYS-16-11060
Record Dates: First submitted 2018-08-02; First posted 2018-09-07 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Stroke, Ischemic; Inflammatory Response; Stroke, Acute
Keywords: TSPO; MRI; PET; Stroke; Brain inflammation
MeSH Terms: conditions — Ischemic Stroke; Stroke; Encephalitis | interventions — Neuroimaging; Magnetic Resonance Imaging; Positron-Emission Tomography; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: Exploratory, prospective, natural history, imaging cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute stroke cohort (Experimental): Acute stroke cohort
  Interventions: Diagnostic Test: Brain Imaging

INTERVENTIONS:
Diagnostic Test: Brain Imaging — The study involves an initial screening visit and 2 study imaging visits at days 15 and 90 after the stroke episode.Patients will undergo:
  1. Two 90-minute brain imaging sessions using Positron Emission Tomography (PET) (involves injection of safe radiotracers which attach to brain immune cell markers TSPOs and light up the inflamed areas in the brain),
  2. Two 45-90 minute Magnetic Resonance Imaging (MRI) scanning sessions (include administration of safe chemical contrast agent Gadolinium),
  3. Physical and neurological examinations (vital signs, assessments of mobility and cognitive functioning),
  4. Blood testing (routine measurements, blood inflammation markers, and genetic testing for TSPO marker).
  Venous cannula will be inserted into the forearm for the duration of the scans.
  Other Names: Magnetic Resonance Imaging (MRI); Positron Emission Tomography (PET-CT)

SUMMARY:
DESIGN: exploratory, prospective, natural history, imaging cohort study

BACKGROUND: Stroke causes a strong inflammatory response in the brain which is thought to contribute to permanent brain damage in stroke patients. To develop new therapies targeting inflammation we need to better understand how inflammation affects the injured brain tissue and how it relates to neurological deficits that directly affect the patients' quality of life.

AIMS: To track the extent and location of inflammation in the brain after stroke over a period of 90 days. The study will explore whether the most inflamed areas in the brain undergo the most damage after stroke and correspond to the cognitive and neurological deficits experienced by stroke patients.

METHODS: The study involves an initial screening visit and 2 study imaging visits at days 15 and 90 after the stroke episode. Patients will undergo:

1. Two 90-minute brain imaging sessions using Positron Emission Tomography (PET) (involves injection of safe radiotracers which attach to brain immune cell markers TSPOs and light up the inflamed areas in the brain),
2. Two 45-90 minute Magnetic Resonance Imaging (MRI) scanning sessions (include administration of safe chemical contrast agent Gadolinium),
3. Physical and neurological examinations (vital signs, assessments of mobility and cognitive functioning),
4. Blood testing (routine measurements, blood inflammation markers, and genetic testing for TSPO marker).

Venous cannula will be inserted into the forearm for the duration of the scans.

POPULATION: 15- 25 patients (recruitment will cease once 15 patients have completed the study)

ELIGIBILITY: Male and female stroke patients, aged 18-85, with a recent (within last 10 days) ischemic stroke of moderate severity, able and willing to provide informed consent

LOCATION: Patients will be recruited at the Charing Cross Hospital, Imperial College Healthcare NHS Trust, and study scans will be performed by Invicro Centre for Imaging Sciences, Hammersmith Hospital

DURATION: 18 months FUNDED BY: Biogen Idec Ltd

DETAILED DESCRIPTION:
Stroke is a leading cause of mortality and serious long-term disability. There is a substantial unmet medical need for new therapies that can improve outcomes in acute stroke.

Experimental and pathologic data suggest that peri-infarct inflammation contributes to secondary injury after brain ischemia and that blocking inflammation could reduce the volume of brain infarction and improve clinical outcome.

In a recently completed phase 2 placebo-controlled clinical trial, the administration of natalizumab (a potent inhibitor of leukocyte transmigration through the blood -brain barrier [BBB]) in the hyperacute phase of ischemic stroke was associated with beneficial effects in measures of functional outcome, but did not affect the rate of infarct volume growth during a 90-day assessment period. This apparent discrepancy between the lack of effect of anti-inflammatory therapy on lesion size and a substantial beneficial effect on functional outcome in ischemic stroke patients has raised further questions about the manifestation of neuroinflammation, its pathophysiological role and its relation to patients' functional outcome in stroke patients.

The purpose of this imaging study is to characterize the subacute and longstanding extent of upregulation of the neuroinflammation marker TSPO on glial cells at two time points after stroke. The study will also explore the correlation of TSPO upregulation with measures of stroke severity and post-stroke functional outcomes.

The objectives of this study are:

* To characterize TSPO glial expression in specific regions of interest defined on correlative brain MRI (ROIs; infarct, peri-infarct, thalamus) in the subacute (day 15+7) and chronic (day 90+/-7) phases after an ischemic stroke;
* To determine the magnitude and variability of TSPO uptake at these ROIs during the assessment period;
* To describe changes in TSPO expression between 15 and 90 days
* To explore the relationship between TSPO uptake, blood and infarct volume, and measures of Wallerian degeneration,
* To characterize post-stroke TSPO glial expression in relation to measures of stroke severity (infarct size, volume and location; NIHSS) and functional outcome (mRS,BI, depression scale, MoCA)
* To characterize post-stroke TSPO glial expression in relation to systemic inflammatory markers in blood

The endpoints that relate to these objectives are:

* PET-derived measures of TSPO radiotracer uptake in the infarct and peri-infarct areas at day 15 and day 90 after a stroke
* PET-derived measures of TSPO radiotracer uptake in ROIs distant from the infarct area (e.g. thalamus, hippocampi, amygdalae and midbrain) at day 15 and day 90 after a stroke
* Correlation of PET-derived measures with clinical and imaging measures of stroke severity (stroke volume, size and NIHSS) and functional outcome (mRS Barthel index, MoCA, depression, ) at day 15 and day 90
* Correlation of infarct volume and MRI measures of white matter tract injury determined from DTI MRI with measures of thalamic TSPO uptake (time-activity curve; measures of mean and max TSPO uptake on summed image sets fromTSPO PET
* Correlation of PET derived measures with inflammatory markers in the blood (e.g. cytokines)

This is an exploratory, prospective, natural history, imaging cohort study. The recruiting site will be Imperial College Healthcare NHS Trust. All study scans will be performed by Invicro, Hammersmith Hospital

Between 15 and 25 subjects, with recruitment ending when 15 participants have completed all study procedures.

Subjects aged 18-85 with a supratentorial ischemic stroke of moderate severity as measured by NIHSS >4 and evidence of infarction on clinical brain scan at time of stroke:

Subjects will participate in this study for approximately 90 days. No treatment will be started as part of the trial

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local subject privacy regulations in accordance with all local and national regulations OR according to the local institutional review board's (IRB's)/ethics committee's (EC's) guidelines OR by another process compliant with applicable national laws and regulations and IRB/EC requirement
2. Aged 18-85 years of age at the time of informed consent
3. Clinical diagnosis of supratentorial acute ischemic stroke within the previous 10 days. Note: An acute brain CT or MRI scan must be available from the patient's history to assess eligibility for the study and be consistent with the diagnosis of acute ischemic stroke.
4. Score of at least 5 points on the NIHSS at Screening.
5. Subjects of childbearing potential (male and female) must be willing and able to practice effective contraception during the study and for 4 weeks after their Day 90 appointment.
6. Negative serum/ urine pregnancy test on all females of childbearing potential within 2 days before each PET study.

Exclusion Criteria:

1. Unable or unwilling to provide informed consent.
2. Presence of acute intracranial hemorrhage on acute brain CT or MRI
3. Inability to comply with study requirements (including implanted pacemaker).
4. Subject has contraindications to undergoing MRI examination (including, but not limited to metal foreign bodies incompatible with MRI exposure, cardiac pacemakers, renal impairment that contraindicates gadolinium etc.) or PET scan.
5. Subject has participated in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with radiation exposure that, when combined with the radiation exposure from the present study, would exceed 10 mSV in addition to the natural background radiation, in the previous 12 months.
6. Other unspecified reasons that, in the opinion of the Investigator make the subject unsuitable for enrollment.
7. Nursing or pregnant females or females planning to become pregnant during study participation.
8. Claustrophobic, unable to hold head continuously still for 90 minutes, or unwilling to undergo PET or MRI imaging and related procedures required for this study.
9. Genetic polymorphism consistent with low TSPO binding affinity (expected in 10% of the population).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute Stroke Cohort: Participants with recent stroke
Period: Overall Study
Arm/Group | Acute Stroke Cohort
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Participants with clinical and radiological acute supratentorial ischaemic stroke within the previous 10 days
Arm/Group | Acute Stroke Cohort
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes in TSPO Radiotracer Uptake Infarct Area
Description: PET-derived measures of TSPO radiotracer uptake in the infarct and peri-infarct areas at day 90 after a stroke (compared with Day 15)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: g/mL
Arm/Group | Acute Stroke Cohort
Number analyzed (Participants) | 3
g/mL | 1.54 (0.39)

2. Primary Outcome: Changes in TSPO Radiotracer Uptake Distant Area
Description: PET-derived measures of TSPO radiotracer uptake in ROIs distant from the infarct area (e.g. thalamus, hippocampi, amygdalae and midbrain) at day 90 after a stroke (compared with Day 15)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: g/mL
Arm/Group | Acute Stroke Cohort
Number analyzed (Participants) | 3
g/mL | 0.89 (0.04)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Acute Stroke Cohort
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT03662750/Prot_SAP_000.pdf